CLINICAL TRIAL: NCT04239651
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) With and Without Internet-Delivered Cognitive Behavior Therapy (iCBT) For the Treatment of Resistant Depression (TRD): Protocol for Patient - Centered Randomized Controlled Pilot Trial
Brief Title: rTMS With and Without iCBT For the Treatment of Resistant Depression (TRD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00094208
Record Dates: First submitted 2019-12-05; First posted 2020-01-27 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-04

CONDITIONS: Depressive Disorder, Treatment-Resistant
Keywords: Repetitive Transcranial Magnetic Stimulation; Internet-Delivered Cognitive Behavior Therapy; Treatment of Resistant Depression; Patient - Centered Randomized Controlled Pilot Trial
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This is a prospective, two-arm randomized controlled trial. 100 patients diagnosed with resistant depression in psychiatric care clinic in Edmonton, Alberta, Canada will be randomized to one of two conditions: (1) enrolment in rTMS sessions alone (2) enrolment in the rTMS sessions plus iCBT.
Who Masked: Outcomes Assessor
Masking Description: Because it will not be possible for participants to be blinded, treatment allocation will be made explicit to them as soon as randomization is concluded. Primary outcome assessors will be blinded to treatment group allocation by not involving them in discussions about study participants and not granting them access to the database which contains the randomization code. After data collection is complete, all data will undergo a blind review for the purposes of finalizing the planned analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enrolment in rTMS sessions alone (Active Comparator): All patients will be scheduled to receive 30 sessions of rTMS treatments over a six-week period as pre-determined by Alberta Health Services' Strategic Clinical Network for Addiction and Mental Health.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Enrolment in iCBT Plus rTMS (Active Comparator): Patients in the rTMS plus iCBT arm of the study, would be assisted to register on the iCBT program (Moodgym) to receive unique login information. They would be assisted to participate in 12 one-hour sessions of iCBT at the clinic prior to receiving rTMS treatments. These in-clinic iCBT sessions would be scheduled in about three days intervals (ideally Tuesdays and Thursdays) so that patients receive two iCBT sessions each week. Patients would also be encouraged to continue with iCBT treatments on their own at home outside the sessions delivered in the clinic.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Other: Internet-Delivered Cognitive Behavior Therapy (iCBT)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — rTMS uses powerful (1.0-2.5 Tesla), focused magnetic field pulses to induce electrical currents in neural tissue noninvasively, via an inductor coil placed against the scalp.
Other: Internet-Delivered Cognitive Behavior Therapy (iCBT) — Cognitive behavioral therapy (CBT) is an evidence-based, structured, intensive, time-limited, symptom-focused form of psychotherapy recommended for the treatment of major depression and anxiety disorders. Internet-delivered CBT (iCBT) is structured CBT delivered via the internet.
  Arms: Enrolment in iCBT Plus rTMS

SUMMARY:
This is a prospective, two-arm randomized controlled trial. 100 patients diagnosed with resistant depression in psychiatric care clinic in Edmonton, Alberta, Canada will be randomized to one of two conditions: (1) enrolment in rTMS sessions alone (2) enrolment in the rTMS sessions plus iCBT. Patients in each group will complete evaluation measures (eg, recovery, general symptomatology and functional outcomes) at baseline, 1 month, 3 months and 6 months. The primary outcome measure would be changes to scores on the Hamilton Depression Rating Scale. Patient service utilization data and clinician-rated measures will also be used to gauge patient progress. Patient data will be analyzed with descriptive statistics, repeated measures and correlational analyses.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE:

Major depression is a severe, disabling, and potentially lethal clinical disorder. While there are a wide variety of pharmaceutical agents available as treatments for major depression, only about half of patients respond to an initial course of antidepressant pharmacotherapy, It has been conservatively estimated that at least 15% of all patients with major depressive disorder remain refractory to any treatment intervention. While a complex relationship exists between disease chronicity and ineffective treatment, clinical evidence suggests that the greater the number of treatment failures, the less likelihood of a good treatment response to subsequent interventions. The reported results of the STAR*D study are the most vivid example of this clinical phenomenon. In that work, there was a progressive likelihood of poorer response with each successive treatment failure. For example, after the first treatment attempt, about 30% of patients remitted. By the time that a patient had experienced definitive treatment failures, the likelihood of achieving remission with the fourth treatment option offered fell below 10%. Taken together, these facts underline the clinical urgency for physicians to identify treatment resistant patients as early as possible so that alternative treatments with proven efficacies may be offered sooner. In turn, this will result in superior treatment outcomes for these treatment resistant patients.

Technology and the Internet have dramatically changed medicine. According to Statistics Canada, 83% of Canadians had Internet access in 2012, and more than 70% use the Internet daily; 62% were smartphone users. E-Mental health refers to the use of computers, Internet, and mobile devices for mental health information and care. E-Mental health applications are now widely available for information, screening, assessment and monitoring, interactive self-management, psychotherapy, and social support. Clinicians should be aware that there are benefits and potential harms to using and recommending e-Mental health applications and that few have good-quality evidence to support effectiveness. Meta-analyses and reviews of computer-based psychological treatment for the treatment of MDD, whether delivered over the Internet or as a stand-alone program, demonstrate convincing support for these treatment modalities. Internet- and computer-delivered cognitive behaviour therapy (iCBT) can also be helpful in relapse prevention.

In 2009, the Canadian Network for Mood and Anxiety Treatments (CANMAT), a not-for-profit scientific and educational organization, published a revision of evidence-based clinical guidelines for the treatment of depressive disorders. CANMAT has updated these guidelines in 2016 to reflect new evidence in the field. Neurostimulation, or neuromodulation, is an expanding area of research and clinical interest, driven in part by the increasing knowledge base on the neurocircuitry of depression. Most of these neurostimulation treatments have been studied and are used in patients with TRD who have failed to respond to standard treatments. However, there is no previous study which has examined the effect of rTMS plus iCBT in comparison to rTMS alone.

Repetitive Transcranial Magnetic Stimulation (rTMS):

rTMS uses powerful (1.0-2.5 Tesla), focused magnetic field pulses to induce electrical currents in neural tissue noninvasively, via an inductor coil placed against the scalp. Therapeutic rTMS is usually delivered by a trained technician or nurse, under physician supervision. Unlike Electroconvulsive Therapy (ECT), no anesthesia is required. The therapeutic mechanism of rTMS is still under investigation, with mechanisms proposed at both cell-molecular and network levels. Repeated rTMS sessions can exert therapeutic effects lasting several months. Clinical trials and naturalistic studies have found maximal effects at 26 to 28 sessions. Clinical experience concurs in suggesting 20 sessions before declaring treatment failure, with extension to 25 to 30 sessions if improvements occur.

More than 30 systematic reviews and meta-analyses have been conducted on rTMS in depression, with most studies involving patients with some degree of treatment resistance (i.e., having failed at least 1 or 2 antidepressant trials). Overall, rTMS is considered a first-line treatment for MDD for patients who have failed at least 1 antidepressant treatment.

Cognitive behavioral therapy (CBT) Psychotherapy:

Cognitive behavioral therapy (CBT) is an evidence-based, structured, intensive, time-limited, symptom-focused form of psychotherapy recommended for the treatment of major depression and anxiety disorders. Internet-delivered CBT (iCBT) is structured CBT delivered via the internet. Cognitive behavioral therapy helps people become aware of how certain negative automatic thoughts, attitudes, expectations, and beliefs contribute to feelings of sadness and anxiety. People undergoing CBT learn how their thinking patterns, which may have developed in the past to deal with difficult or painful experiences, can be identified and changed to reduce unhappiness.

Barriers to face-to-face conventional ways for treatment include stigmas around people seeking help in person, geography (distance from health care professional), time, and cost. Increasingly, there is a desire to pursue internet delivery as an option to increase access to treatment.

Internet-delivered CBT (iCBT) consists of structured modules with clearly defined goals, and is delivered via the internet. Although there are many types of iCBT programs, each are goal-oriented sessions that typically consist of 8 to 12 modules and can be guided or unguided. Internet-delivered CBT programs are made available by computer, smartphone, or tablet, for a fee. With unguided iCBT, patients are informed of a website through which they can participate in an online self-directed program. Guided iCBT involves support from a regulated health professional (e.g., social worker, psychologist, psychotherapist, occupational therapist, nurse, or physician). In guided iCBT, people complete modules and communicate (via email, text messages, or telephone calls) their progress to a regulated health professional.

OBJECTIVES A goal of the project is to evaluate the feasibility of implementing rTMS plus iCBT for treatment of patients diagnosed with TRD. Another goal of the project is to assess the initial comparative clinical effectiveness of rTMS treatments when used with and without iCBT.

Because of the limited availability of data in this specific area, another goal of the study is to generate effect size data for these interventions which will help in sample size and power calculations for a full randomized clinical trial. The patient's outcomes are organized according to: recovery variables (eg, recovery and stigma), functional variables (quality of life and employment), symptom variables (psychological symptoms and general outcomes) and other outcomes will be service variables (eg, heath service utilization, cost and satisfaction).

METHODS:

This study will be a prospective, parallel design, two-arm, rater-blinded Randomized Controlled Trial (RCT) with a recruitment period of 12 months and applying active treatment for 6 weeks and an observation period of 6 months for each participant. The research will be carried out in an Addiction and Mental Health clinic in a large, socio-demographically diverse city in Western Canada (Edmonton, Alberta).

INTERVENTIONS Patients would be randomly assigned to receive either rTMS alone or rTMSplus iCBT Patients in both arms of the study will be assigned to an introductory visit to introduce the rTMS system to them and explain the procedure which will be carried out in each visit. All patients will be scheduled to receive 30 sessions of rTMS treatments over a six-week period as pre-determined by Alberta Health Services' Strategic Clinical Network for Addiction and Mental Health. In addition, patients in the rTMS plus iCBT arm of the study, would be assisted to register on the iCBT program (MoodGym) to receive unique login information. To reduce in-person contact due to COVID-19 protocols, patients would be remotely assisted via phone to participate in 12 one-hour sessions of iCBT at the clinic prior to receiving rTMS treatments. These iCBT sessions would be scheduled in about three days intervals (ideally Tuesdays and Thursdays) so that patients receive two iCBT sessions each week. Patients would also be encouraged to continue with iCBT treatments beyond the scheduled sessions.

All patients will be followed up for 6 months and would be encouraged to continue to receive whatever community clinic/ program treatments or supports are part of their usual care.

HYPOTHESIS The investigators hypothesize that patients enrolled in the rTMS plus iCBT treatment arm of the study will achieve superior outcomes compared with patients enrolled in the rTMS alone arm of the study on each outcome measure used.

SAMPLE SIZE The study will therefore be limited to a sample size of 100, with about 50 patients recruited into each arm of the study. Patients transitioning from resistance of the pharmacological treatment are vulnerable to severe depressive attacks, and it can reasonably be expected that only a small number of eligible participants will enroll in and complete the study.

RANDOMIZATION AND BLINDING Randomization will be stratified by using permuted blocks to ensure balance (1:1) between the two follow-up treatment groups. The randomization codes will be transmitted by an independent statistician via text message directly to a researcher's password-protected phone line with a secure online backup. This will commence as soon as participants sign the consent forms.

Because it will not be possible for participants to be blinded, treatment allocation will be made explicit to them as soon as randomization is concluded. Primary outcome assessors will be blinded to treatment group allocation by not involving them in discussions about study participants and not granting them access to the database which contains the randomization code. After data collection is complete, all data will undergo a blind review for the purposes of finalizing the planned analysis.

FOLLOW-UP ASSESSMENT At 1, 3 and 6 months, a blinded researcher will contact all study participants and assist them to complete a range of assessment tools relating to the primary and secondary outcome measures. They will be offered the opportunity to complete the assessments face to face or over the phone. At 6 months, data related to each person's clinic/ programme attendance rates and utilization of health services will be compiled from administrative records by the blinded researcher.

PATIENT AND PUBLIC INVOLVEMENT This study was designed to address the clinical urgency to identify and respond to early evidence of treatment resistance using treatments that have proven efficacy in these more difficult-to-treat psychiatric patients. The study is designed as patient-oriented research with the active involvement of a patient representative who will be a coauthor of the study protocol. The randomized trial offers patients the opportunity to provide feedback regarding the burden of the intervention through a focused group workshop involving a cross section of patients in the two arms of the study.

ETHICS AND DISSEMINATION The study will be conducted in accordance with the Declaration of Helsinki (Hong Kong Amendment) and Good Clinical Practice (Canadian Guidelines). Written informed consent will be obtained from each participant. The study results, expected 18 months after commencement of recruitment, will be disseminated at several levels, including patients, practitioners, academics/researchers, and healthcare organizations.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-60 years
* Suffering from a major depressive episode based on Diagnostic and Statistical manual (DSM) 5 criteria and having failed two or more standard antidepressant treatments during the current episode.
* Hamilton Depression Rating Scale (17-HAM-D) score of 21 or more
* Participant may be on psychotropic medications including antidepressants, antipsychotics, benzodiazepines and anticonvulsants
* Able and willing to provide informed consent.

Exclusion Criteria:

* Diagnosis with the following conditions (current unless otherwise stated):

  * Have a neurological disorder, including a history of seizures, cerebrovascular disease, primary or secondary tumors in central nervous system, stroke, cerebral aneurysm or movement disorder or any lifetime history of loss of consciousness due to head injury.
  * Any current Axis 1 psychotic disorder (including substance-induced psychosis, psychotic disorder due to a medical condition, or major depression with psychotic features), as defined by the MINI (Mini International Neuropsychiatric Interview; English Version 7.0.0 for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5); Copyright 1992---2014 Sheehan DV) at the screening visit.
  * Any lifetime Axis 1 psychotic disorder (excluding substance-induced psychosis, or psychotic disorder due to a medical condition), or as defined by the MINI at the screening visit.
  * Any current Axis II personality disorder that would interfere in the participation of the study as determined or might affect cognition and ability to meaningfully participate. In addition to mental retardation identified through medical history or in the opinion of the investigator.
  * Have a current amnestic disorder, dementia, or delirium as defined by Montreal Cognitive Assessment of less than or equal to 16 or any other neurological or mental disease that might affect cognition or the ability to meaningfully participate in cognitive behavioral therapy (CBT).
  * Any illicit substance use as determined by positive toxicology screen for drugs of abuse; or alcohol and/or substance abuse or dependence within the past 3 months (90 days) as determined by the MINI at the screening visit
* Treatment histories including prior treatment with TMS.
* Have active suicidal intent or plan as defined by a positive answer to questions 4 and/or 5 on the Columbia-Suicide Severity Rating Scale (CSSRS): Screening version; or more than one suicide attempt in lifetime; or a suicide attempt in the past twelve months; or in the Investigator's opinion, is likely to attempt suicide within the next six months.
* Participation in any drug or device clinical trial in the six weeks (42 days) prior to the screening visit and/or participation in another clinical trial for the duration of the study.
* Presence of any other condition or circumstance that, in the opinion of the investigator, has the potential to prevent study completion and/or to have a confounding effect on outcome assessments.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
The Hamilton Depression Rating Scale. | 6 months
  The scale contains 17 variables. Some are defined in terms of a series of categories of increasing intensity, while others are defined by a number of equal-valued terms. The form on which ratings are recorded also includes: four :Diurnal variation, de- realization, paranoid symptoms, obsessional symptoms.score Range of its score is from 0-54. from 0-6 means no depression.
  7-17: mild depression 18-24:moderate depression 24 and more: Severe depression

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptomatology Self Report-16. | 6 months
  To assess depression as a symptom variable. Total scores range from 0 to 27 and high score means the worse outcome .The total score is obtained by adding the scores for each of the nine symptom domains of the DSM-IV MDD criteria: depressed mood, loss of interest or pleasure, concentration/decision making, self-outlook, suicidal ideation, energy/fatiguability, sleep, weight/appetite change, and psychomotor changes.
Columbia Suicide Severity Rating Scale. | 6 months
  To assess suicidal ideation as symptom variable. Suicidal Ideation Score: The maximum suicidal ideation category (1-5 on the C- SSRS) present at the assessment. Assign a score of 0 if no ideation is present.
Young Mania Rating Scale. | 6 months
  To assess mania as a symptom variable.There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. These four items are given twice the weight of the others to compensate for poor cooperation from severely ill patients. There are well described anchor points for each grade of severity. The authors encourage the use of whole or half point ratings once experience with the scale is acquired. Typical YMRS baseline scores can vary a lot. They depend on the patients' clinical features such as mania (YMRS = 12), depression (YMRS = 3), or euthymia (YMRS = 2). Sometimes a clinical study entry requirement of YMRS > 20 generates a mean YMRS baseline of about 30. Strengths of the YMRS include its brevity, widely accepted use, and ease of administration. The usefulness of the scale is limited in populations with diagnoses other than mania.
Frequency, Intensity, and Burden of Side Effects Ratings *Edited for rTMS | 6 months
  To assess side effects as a functional variable. A patient self-report used to quantify the overall side effect burden. Used in combination with the PRISE. Rated for the last 7 days. Each item uses a 7-point Likert-type scale rated from 0 (i.e. no side effects) to 6 (i.e. intolerable). 3 global ratings encompass all side effects to study treatment experienced over the past week. One item rates frequency, another rating the intensity of side effects encountered in the prior week that the participant believes were due to the antidepressant treatment, and the third asks participants to estimate the overall burden or degree of interference in day-to-day activities and functioning due to the side effects.
Patient Rated Inventory of Side Effects. | 6 months
  To assess side effects as a functional variable. A patient self-report used to qualify side effects by identifying and evaluating the tolerability of each symptoms. Used in combination with the FIBSER. Rated for the last 7 days. 7 item assessment of the side effects in the following symptom domains; Gastrointestinal, Heart, Skin, Nervous System, Eyes/Ears, Genital/Urinary, Sleep, Sexual Functioning, and Other. Each domain has multiple symptoms which can be endorsed. For each domain the patient rates whether or not the symptoms are tolerable or distressing.
World Health Organization Disability Assessment 2.0 | 6 months
  To assess disability as a functional variable.The scoring has three steps:
  Step 1 - Summing of recoded item scores within each domain. Step 2 - Summing of all six domain scores. Step 3 - Converting the summary score into a metric ranging from 0 to 100 (where 0 = no disability; 100 = full disability).
(The EuroQol-5 Dimension Assessment). | 6 months
  To assess the quality of life as a functional variable.
  Each of the five dimensions comprising the EQ-5D descriptive system is divided into five levels of perceived problems:
  LEVEL 1: indicating no problem LEVEL 2: indicating slight problems LEVEL 3: indicating moderate problems LEVEL 4: indicating severe problems LEVEL 5: indicating unable to/extreme problems A unique health state is defined by combining one level from each of the five dimensions.
Patient Satisfaction/ Community Service Experience Survey | 3 months
  To assess patient satisfaction with service as a service variable.Identify survey questions that receive low scores and prioritize improving those areas (i.e., connect them to investigators strategic goals or propose them as an area of focus for the Board). Benchmark results against:
  * The previous survey results
  * Investigators peers
  * Industry standard
  * Best practices
  * "Bright spots" in primary care

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Agyapong, MD,Ph.D, Principal Investigator — Division of Community Psychiatry, University of Alberta
Locations (1):
- Edmonton Mental Health Clinic, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abou El-Magd RM, Obuobi-Donkor G, Adu MK, Lachowski C, Duddumpudi S, Lawal MA, Sapara AO, Achor M, Kouzehgaran M, Hegde R, Chew C, Mach M, Daubert S, Urichuk L, Snaterse M, Surood S, Li D, Greenshaw A, Agyapong VIO. Repetitive Transcranial Magnetic Stimulation With and Without Internet-Delivered Cognitive-Behavioral Therapy for the Treatment of Resistant Depression: Protocol for Patient-Centered Randomized Controlled Pilot Trial. JMIR Res Protoc. 2020 Oct 27;9(10):e18843. doi: 10.2196/18843. PMID 33107835